CLINICAL TRIAL: NCT03971825
Title: A Phase 1, Randomized, 3-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of CC-92252 in Healthy Adult Subjects and Adult Subjects With Psoriasis.
Brief Title: A Safety Study of CC-92252 in Healthy Adult Subjects and Adult Subjects With Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not meet progression criteria
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-92252-CP-001; U1111-1229-5867 (Registry Identifier: WHO); 2018-001050-10 (EudraCT Number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers; Psoriasis
Keywords: Psoriasis; Healthy Volunteer; Safety; CC-92252
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Administration of CC-92252 and Placebo in Healthy Subjects (Experimental): Part 1 of the study will be conducted as a single ascending dose study, each cohort will consist of 9 subjects. Part 2 of the study will be conducted as a multiple ascending dose study, each cohort will consist of 8 subjects. In part 3, subjects with psoriasis will receive CC-92252 or placebo for up to 12 weeks.
  Interventions: Drug: CC-92252; Other: Placebo
- Administration of CC-92252 and Placebo in Psoriasis subjects (Experimental): Part 1 of the study will be conducted as a single ascending dose study, each cohort will consist of 9 subjects. Part 2 of the study will be conducted as a multiple ascending dose study, each cohort will consist of 8 subjects. In part 3, subjects with psoris will receive CC-92252 or placebo for up to 12 weeks.
  Interventions: Drug: CC-92252; Other: Placebo

INTERVENTIONS:
Drug: CC-92252 — CC-92252
Other: Placebo — Placebo

SUMMARY:
This is a phase 1, randomized, single-center, 3-part, study to assess the safety, tolerability, PK, and PD, of single and multiple doses of CC-92252 in healthy adult subjects and multiple doses of CC-92252 in adult subjects with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

Part 1, Part 2, and Part 3

1. Subject is ≥ 18 and ≤ 55 years (Part 1 and Part 2) and age is ≥ 18 and ≤ 60 years (Part 3) of age at the time of signing the ICF.
2. Subject has provided informed consent prior to initiation of any study specific activities/procedures
3. Subject has a body mass index (BMI) ≥ 18 and ≤ 30 kg/m2 (Part 1 and Part 2) and BMI ≥ 18 and ≤ 33 kg/m2 (Part 3), at screening.
4. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator.

   Applicable to Part 3 only
5. Subject has a clinical diagnosis of stable plaque-type PsO at least 6 months prior to screening, defined as:

   BSA ≥ 5% (at both screening and baseline), and sPGA score ≥ 3 (at both screening and baseline)
6. Must have at least two plaques, at least 3 x 3 centimeters (cm) in diameter. One plaque will be used for punch biopsy and the other for Target Plaque Severity Score (TPSS) evaluation.
7. Must be in generally good health (except for PsO) as judged by the Investigator
8. No prior exposure to systemic treatments or biologics for the treatment of psoriasis

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

Part 1, Part 2, and Part 3

1. Subject has any significant medical condition that would prevent the subject from participating in the study.

   a. Part 3 only: This exclusion does not apply to plaque psoriasis
2. History or presence of cancer
3. Presence of pre-cancerous conditions
4. History or presence of a systemic infection or any potentially opportunistic infections
5. Subject has any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
6. Subject has any condition that confounds the ability to interpret data from the study
7. Subject is pregnant or breastfeeding
8. Part 1 and Part 2 only: Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer)
9. Part 1 and Part 2 only: Subject has used any prescribed systemic or topical medication within 30 days prior to the first dose administration.
10. Part 1 and Part 2 only: Subject has used any non-prescribed systemic or topical medication within 14 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to and documented by the Investigator and Sponsor's Medical Monitor.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs
12. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years before the first dose administration, or positive alcohol screen
13. Subject is known to have a history of hepatitis B and/or hepatitis C, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening Note: Subjects who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation
14. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported)
15. Vaccination within 30 days prior to the first dose administration or subject has plans to receive a vaccination during the course of the study
16. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to the first dose administration or is planning to receive immunization with a live or live attenuated vaccine for 2 months following the last dose administration
17. Subject has a positive QuantiFERON®-TB Gold (or equivalent) TB test at screening or 2 successive indeterminate QuantiFERON®-TB Gold (or equivalent) TB tests at screening
18. Subject has a history of incompletely treated Mycobacterium tuberculosis (TB) infection
19. Topical therapy within 2 weeks of randomization (including, but not limited to, topical corticosteroids, retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol). Use of phototherapy within 4 weeks prior to first dose administration.
20. Prolonged sun exposure or use of tanning booths Applicable to Part 3 only
21. Presence of non-plaque psoriasis
22. Subject has psoriasis flare within 4 weeks before screening
23. Presence of dermatological diseases other than plaque psoriasis
24. Presence of Psoriatic Arthritis
25. Use of topical therapy for psoriasis within 14 days of first dosing (including but not limited to corticosteroids, retinoids, vitamin D analog, calcineurin inhibitors, salicylic acid) Exceptions: low potency topical corticosteroids will be allowed as background therapy for treatment of psoriatic lesions of the face, axillae and groin in accordance with the manufacturers' suggested usage; subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions; Eucerin® cream (the standard emollient for this study; or equivalent) will also be permitted for body lesions only. Subjects must not use these treatments within 24 hours prior to each clinic visit.
26. Use of systemic therapy for psoriasis within 30 days of first dose administration
27. Use of phototherapy for psoriasis within 30 days of first dose administration
28. Use of systemic biologic treatment within 24 weeks of first dose administration
29. Exposure to an immunosuppressive or immunomodulatory drug within 30 days of first dose administration, or five half-lives of the drug (whichever is longer)
30. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse event

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Up to 16 weeks
  Observed maximum serum concentration
Pharmacokinetics - AUC0-t | Up to 16 weeks
  Area under the serum concentration-time curve calculated from time zero to the last measured time point
Pharmacokinetics - AUC0-∞ | Up to 16 weeks
  The area under the curve extrapolated to infinity, calculated using the observed value of the last non-zero concentration
Pharmacokinetics - Tmax | Up to 16 weeks
  Time to Cmax
Pharmacokinetics - t1/2z | UP to 16 weeks
  Terminal elimination half-life
Pharmacokinetics - CL/F | Up to 16 weeks
  Apparent clearance of drug from serum after subcutaneous dosing administration
Pharmacokinetics - CL | Up to 16 weeks
  clearance of drug from serum after IV dosing
Pharmacokinetics - Vz/F | Up to 16 weeks
  Apparent volume of distribution during the terminal phase
Pharmacokinetics - Vz | Up to 16 weeks
  Apparent volume of distribution during the terminal phase
Anti-drug Antibody Immunogenicity Anti-drug antibody | Up to 16 weeks
  Evaluation of anti-CC-92252 antibody formation
Assessment of Pharmacodynamic biomarkers | UP to 24 weeks
  Change in lymphocyte counts

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramirez-Valle, MD, PhD, Study Director — Celgene
Locations (1):
- Charite Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/